CLINICAL TRIAL: NCT04509401
Title: The Neurobehavioral and Biochemical Effects of High Dose of Vitamin B6 With Magnesium in Children With Autism Spectrum Disorder: A Randomized, Double-Blind, Placebo Controlled Study
Brief Title: Effects of High Dose of Vitamin B6 With Magnesium in Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Fatema Ershad, Principal Investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BSMMU/2019/12342
Record Dates: First submitted 2020-07-29; First posted 2020-08-12 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: ASD
Keywords: Vitamin B6; Magnesium; Homovanillic acid; ADCL; ASD
MeSH Terms: interventions — Vitamin B 6; Magnesium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Active Comparator): High dose of Vitamin B6 with Magnesium. Vitamin B6 will be given orally 150 mg for ages 2-3 years, 200 mg for ages 4-6 years,300 mg for ages 7-8 years and Magnesium will be given orally 50 mg for 2-3 years, 100 mg for ages 7-8 years for three months.
  Interventions: Drug: Vitamin B 6 with Magnesium
- Control (Placebo Comparator): Control group will receive oral placebo in the same manner, schedule and time frame.
  Interventions: Drug: placebo of vitamin B6 and magnesium

INTERVENTIONS:
Drug: Vitamin B 6 with Magnesium — Patients of intervention group will receive high dose of vitamin B6 with magnesium. This group will receive high dose of vitamin B6 with magnesium orally for 12 weeks.
  Arms: Interventional
Drug: placebo of vitamin B6 and magnesium — Patients of control group will receive oral placebo tablet in the same manner, schedule for 12 weeks.
  Arms: Control

SUMMARY:
Title:

The Neurobehavioral and Biochemical Effects of High Does of Vitamin B6 with Magnesium in Children with Autism spectrum Disorder: A Randomized, Double-Blind, Placebo Controlled Study.

Purpose of the Study:

This study aims to examine the effect of higher doses of vitamin B6-magnesium combination in modification of urinary homovanillic acid excretion and improving behavioral sign symptoms in a newly diagnosed autistic children.

Method:

This study will be a randomized,double blind placebo controlled trial to assess the effects of high dose of vitamin B6 with magnesium upon autistic children. This study will be conducted in the Department of Pharmacology and Institute of Pediatric Neurodisorder and Autism (IPNA) in between July 2019 to July 2020. A total 66 newly diagnosed autistic children will be selected according to inclusion and exclusion criteria. The patients will be divided randomly into 2 groups: Intervention group and Control group. Intervention group will consist of 33 patients who will receive vitamin B6-magnesium along with standard care of treatment for three months. Vitamin B6 will be given 150 mg for ages 2-3 years, 200 mg for ages 4-6 years, 300 mg for ages 7-8 years and Magnesium will be given 50 mg 2-4 years, 100 mg for ages 4-8 years. Control group consist of 33 patients who will receive placebo in the same manners along with standard care of treatment for three months. To see the effects of Vitamin B6 and Magnesium, Autism Spectrum Disorder would be assessed by Autism Diagnostic Checklist (ADCL) at baseline and three months after intervention. Urinary homovanillic acid level would also be performed at baseline and three months after intervention.

Ethical consideration:

The study will follow the principles of the Declaration of Helsinki and of the World Medical Assembly. Parents of the patient will be informed about the study in easy language and then informed written consent will be taken. This study has no potential risk to the patients. Confidentiality will be strictly maintained.

DETAILED DESCRIPTION:
Autism spectrum Disorder is a complex neuro- developmental, incurable disease with lifelong impacts.Epidemiological studies have shown a rapid increase in the prevalence of ASD throughout the world including Bangladesh. The World Health Organization (WHO) estimated every 1 in 160 children has an autism spectrum disorder. Various environmental, genetic ,biochemical, metabolic factors are presumed to be involved in the etiology of ASD. Researchers found Vitamin B6 with Magnesium has the potential effects to alleviate the core symptoms of autism. A possible association higher doses of vitamin B6-Magnesium supplementation may reduce biochemical abnormalities e.g. reduction of urinary excretion of homovanillic acid and improve neurobehavioral symptoms.Therefore the present study has been designed to assess the effects of high dose of vitamin B6 with magnesium along with standard care of treatment upon ASD patients. The study would be randomized, double blind placebo controlled trial to be conducted in the Department of Pharmacology and the Institute of Pediatric Neurodisoder and Autism(IPNA), BSMMU in between July 2019 to July 2020. A total 66 newly diagnosed ASD patients will be selected according to inclusion and exclusion criteria. The patients will be divided randomly into 2 groups: intervention and control. Intervention group would consist of 33 patients who wlill receive high dose of vitamin B6 with magnesium orally for three months. Vitamin B6 will be given 50 mg for 2- 3 years, 200 mg for ages 4-6 years, 300 mg for ages 7-8 years and Magnesium will be given 50 mg for 2-3 years, 100 mg for ages 4-8 years. Control group would also consist of 33 patients who will receive placebo in the same manners along with standard care of treatment for three months. Comparison between the two groups will be performed through urinary homovanillic acid estimation at baseline and three months after the intervention. Neurobehavioral status will be assess by Autism Diagnostic Checklist (ADCL) at baseline and after three months of intervention. Data would be analyzed by Scientific Package for Social Science and represented by tables and figures as applicable. Significance level would be set at 0.05, 0.01 and 0.001. Patients data will be recorded in a predetermined data sheet. Parents of the patient will be informed about the study in easy language and then written informed consent will be taken.This study has no potential risk to the patients.

ELIGIBILITY:
Inclusion Criteria: Newly diagnosed patients of Autism Spectrum Disorder Co-morbid neurological disorder like irritability, hyperactivity with ASD

-

Exclusion Criteria: Epilepsy

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2020-01-11 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
To measure the urinary homovanillic acid Conc in µgm/mg of creatinine in Vitamin B6 with magnesium treated autistic children pre and post supplementation of Vitamin B6 and Magnesium. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fatema Ershad, MBBS, Principal Investigator — BSMMU (Recruiting)
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No